CLINICAL TRIAL: NCT04448431
Title: A Randomised, Double-blind, Parallel-group, Active Controlled Study Evaluating the Efficacy of Vortioxetine Versus Desvenlafaxine in Adult Patients Suffering From Major Depressive Disorder With Partial Response to SSRI Treatment
Brief Title: Comparison of Vortioxetine and Desvenlafaxine in Adult Patients Suffering From Depression
Acronym: VIVRE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18498A
Record Dates: First submitted 2020-06-23; First posted 2020-06-25 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Vortioxetine; Desvenlafaxine Succinate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vortioxetine (Experimental): 8 weeks treatment
  Interventions: Drug: Vortioxetine
- Desvenlafaxine (Active Comparator): 8 weeks treatment
  Interventions: Drug: Desvenlafaxine

INTERVENTIONS:
Drug: Vortioxetine — 10 or 20 mg/day, capsules, orally
  Arms: Vortioxetine
Drug: Desvenlafaxine — 50 mg/day capsules, orally
  Arms: Desvenlafaxine

SUMMARY:
The purpose of this study is to compare the efficacy of vortioxetine versus desvenlafaxine after 8 weeks of treatment in patients that have tried one available treatment without getting the full benefit

DETAILED DESCRIPTION:
The study will consist of a screening period of up to 14 days before the Baseline Visit, followed by an 8-week Treatment Period with vortioxetine or desvenlafaxine. A Safety Follow-up Visit will be performed approximately 4 weeks after the Primary Outcome/Withdrawal Visit.

At Baseline, patients will be equally randomised (1:1) to 1 of the 2 treatment groups for an 8-week, double-blind Treatment Period.

ELIGIBILITY:
Inclusion Criteria:

* The patient has a primary diagnosis of single or recurrent MDD, diagnosed according to DSM-5®. The current MDE must be confirmed using the Mini International Neuropsychiatric Interview (MINI).
* The patient has a MADRS total score ≥24 at screening and baseline.
* The patient has had the current MDE for ≥3 months and < 12 months.
* The patient has been treated with an SSRI as monotherapy (citalopram, escitalopram, paroxetine, sertraline) for at least 6 weeks at licensed dose for the current MDE with a partial response and is a candidate for a switch in the investigator's opinion.
* The patient wants to switch antidepressant treatment.

Exclusion Criteria:

* The patient has any other disorder for which the treatment takes priority over treatment of MDD or is likely to interfere with study treatment or impair treatment compliance.

Other in- and exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 605 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2022-01-06 (Actual); Study Completion 2022-02-04 (Actual)

PRIMARY OUTCOMES:
Change in Montgomery and Åsberg Depression Rating Scale (MADRS) total score | From baseline to Week 8
  The Montgomery and Åsberg Depression Rating Scale (MADRS) is a 10-item rating scale designed to assess the severity of the symptoms in depressive illness and to be sensitive to treatment effects. Symptoms are rated on a 7-point scale from 0 (no symptom) to 6 (severe symptom). The total score of the 10 items ranges from 0 to 60, with higher values indicating worse outcome.

SECONDARY OUTCOMES:
Remission (defined as a MADRS total score =<10) | At Week 8
  The Montgomery and Åsberg Depression Rating Scale (MADRS) is a 10-item rating scale designed to assess the severity of the symptoms in depressive illness and to be sensitive to treatment effects. Symptoms are rated on a 7-point scale from 0 (no symptom) to 6 (severe symptom). The total score of the 10 items ranges from 0 to 60, with higher values indicating worse outcome.
Response (defined as a => 50% decrease from baseline in MADRS total score) | At Week 8
  The Montgomery and Åsberg Depression Rating Scale (MADRS) is a 10-item rating scale designed to assess the severity of the symptoms in depressive illness and to be sensitive to treatment effects. Symptoms are rated on a 7-point scale from 0 (no symptom) to 6 (severe symptom). The total score of the 10 items ranges from 0 to 60, with higher values indicating worse outcome.
Change in MADRS anhedonia factor score | From baseline to Week 8
  (based on items 1(apparent sadness),2 (reported sadness),6 (concentration difficulties),7 (lassitude),8 (inability to feel))
Change in Digital Symbol Substitution Test (DSST) total score | From baseline to Week 8
  DSST assesses psychomotor speed of performance requiring visual perception, spatial decision-making, and motor skills. It consists of 133 digits and requires the patient to substitute each digit with a simple symbol in a 90-s period. Each correct symbol is counted, and the total score ranges from 0 (< normal functioning) to 133 (> normal functioning).
The proportion number of Hard Choice/number of High Reward trials and number of Low choice/number of Low Reward trials when performing the Effort- Expenditure for Rewards Task (EEfRT) | From baseline to Week 8
  The EEfRT is a computerized task which measures reward motivation in which participants are presented with a series of repeated trials during which they choose between performing a ''hard-task'' or an ''easy-task'' in order to earn varying amounts of monetary rewards.
Change in Clinical Global Impression - Severity of Illness (CGI-S) score | from baseline to Week 8
  The CGI-S scale measures the severity of psychiatric symptoms on a 7-point scale from 1-7. The scores indicated the following: 1 = normal, not at all ill; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; 7 = among the most extremely ill participants. The score ranged from 1-7, where 1 indicated absence of symptoms and higher score indicated greater severity of symptoms.
Clinical Global Impression Scale- Global Improvement (CGI-I) score | at Day 7,28,56
  The Clinical Global Impression - global improvement CGI-I provides the clinician's impression of the patient's improvement (or worsening). The clinician assesses the patient's condition relative to a baseline on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse)
Change in Functioning Assessment Short Test (FAST) total score | From baseline to Week 8
  The FAST is a valid and reliable instrument, easy to apply which requires a short period of time to administer. Evaluates functioning taking into account the last 15 days. It was developed for the clinical evaluation of the main difficulties presented by psychiatric patients, and has been validated in several languages for patients with bipolar disorder. The FAST scale consists of 24 items which allow the assessment of six specific areas of functioning: autonomy, occupational functioning, cognitive functioning, financial issues, interpersonal relationships and leisure time
Change in FAST sub-domain scores | From baseline to Week 8
  The FAST is a clinician-rated scale designed to assess difficulty in functioning. The FAST consists of 24 items in 6 specific areas of functioning: autonomy, occupational functioning, cognitive functioning, financial issues, interpersonal relationships, leisure time. Each item is rated on a 4-point scale from 0 (no difficulty) to 3 (severe difficulty). The items are summed to yield a total score ranging from 0 to 72 with higher scores reflecting more serious difficulties.
Change in Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) total score | From baseline to Week 8
  The original Q-LES-Q is a patient self-rated scale designed to measure the degree of enjoyment and satisfaction experienced by patients in various areas of daily life. It consists of 93 items to measure: physical health, feelings, work, household duties, school, leisure time activities, social relations, and general activities. Each item is rated on a 5-point scale ranging from 1 (very poor) to 5 (very good)
Change in Q-LES-Q work subscale | From baseline to Week 8
  The original Q-LES-Q is a patient self-rated scale designed to measure the degree of enjoyment and satisfaction experienced by patients in various areas of daily life. It consists of 93 items to measure: physical health, feelings, work, household duties, school, leisure time activities, social relations, and general activities. Each item is rated on a 5-point scale ranging from 1 (very poor) to 5 (very good)
Change in Q-LES-Q household duties subscale | From baseline to Week 8
  The original Q-LES-Q is a patient self-rated scale designed to measure the degree of enjoyment and satisfaction experienced by patients in various areas of daily life. It consists of 93 items to measure: physical health, feelings, work, household duties, school, leisure time activities, social relations, and general activities. Each item is rated on a 5-point scale ranging from 1 (very poor) to 5 (very good)
Change in Q-LES-Q school/course subscale | From baseline to Week 8
  The original Q-LES-Q is a patient self-rated scale designed to measure the degree of enjoyment and satisfaction experienced by patients in various areas of daily life. It consists of 93 items to measure: physical health, feelings, work, household duties, school, leisure time activities, social relations, and general activities. Each item is rated on a 5-point scale ranging from 1 (very poor) to 5 (very good)
Change in Q-LES-Q leisure time activities subscale | From baseline to Week 8
  The original Q-LES-Q is a patient self-rated scale designed to measure the degree of enjoyment and satisfaction experienced by patients in various areas of daily life. It consists of 93 items to measure: physical health, feelings, work, household duties, school, leisure time activities, social relations, and general activities. Each item is rated on a 5-point scale ranging from 1 (very poor) to 5 (very good)
Change in Q-LES-Q social relations subscale | From baseline to Week 8
  The original Q-LES-Q is a patient self-rated scale designed to measure the degree of enjoyment and satisfaction experienced by patients in various areas of daily life. It consists of 93 items to measure: physical health, feelings, work, household duties, school, leisure time activities, social relations, and general activities. Each item is rated on a 5-point scale ranging from 1 (very poor) to 5 (very good)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (80):
- Argentina (14):
  - Clinica Privada Banfield, Banfield, Buenos Aires
  - Cenydet-Centro Neurobiologico Y De Estres Traumatico-Biopsychomedical Research Group Srl, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Fundacion para el Estudio y Tratamiento de las enfermedades mentales FETEM, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - INAPsi (Instituto Nacional de Psicopatologia), Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Clinica Privada De Salud Mental Santa Teresa De Avila, La Plata, Buenos Aires
  - Instituto De Neurociencias San Agustin SA, La Plata, Buenos Aires
  - Sanatorio Prof. Leon S. Morra S.A., Córdoba, Providencia de Cordo
  - CIAP (Centro de Investigacion y Asistencia en Psiquiatria), Rosario, Santa Fe Province
  - CINME (Centro de Investigaciones Metabolicas de Buenos Aires), Buenos Aires
  - CEN (Centro Especializado Neurociencias), Córdoba
  - Instituto Modelo de Neurologia Fundacion Lennox, Córdoba
  - Instituto Medico DAMIC - Fundacion Rusculleda, Córdoba
  - Centro De Asistencia E Investigacion En Neurociencias CENAIN, Mendoza
  - Resolution Psicopharmacology Research Institute, Mendoza
- Belgium (3):
  - Algemeen Ziekenhuis St. Lucas-St. Jozef, Bruges
  - SINAPS - University Antwerpe- Psychiatrisch Ziekenhuis Duffel, Duffel
  - Cliniques De Mont-Godinne, Yvoir
- Bulgaria (6):
  - MHAT Dr. Hristo Stambolski, Kazanlak
  - UMHAT Sv. Ivan Rilski EAD, Plovdiv
  - Center For Mental Health-Rousse, Rousse
  - MC Complete Medical Solutions, Samokov
  - Centre for Mental Health- Sofia, Sofia
  - Diagnostic Consultative Center Mladost-M Varna OOD, Varna
- Czechia (9):
  - Clintrial s.r.o., Prague, Prague 10
  - Dr.Jan Holan MD, Office of, Brno
  - Meditrine s.r.o. - Psychiatricka Ambulance, Lecebne Centrum, Havířov
  - Clinline services s.r.o., Hostivice
  - Neuropsychiatrie HK, s.r.o., Hradec Králové
  - National Institute of Mental Health, Klecany
  - Psychiatricka Ambulance, Kutná Hora
  - A-Shine s.r.o., Pilsen
  - Institut neuropsychiatricke pece, Prague
- Marienthali Kliinik, Tallinn, Estonia
- Latvia (3):
  - Psihiatrijas Centrs, Liepāja, Liepajas Rajons
  - Riga Centre Of Psychiatry And Addiction Disorders, Riga
  - Sigulda Hospital Outpatient Clinic, Sigulda
- Mexico (3):
  - CRI Centro Regiomontano de Investigacion SC, Monterrey, Nuevo León
  - Medical Care and Research S.A. de C.V., Mérida, Yucatán
  - Health Pharma Professional Research S.A. de C.V., Mexico City
- Russia (15):
  - Region Specialized Psychiatric Hospital No.2, Stavropol Region, Kochubeev District
  - Leningrad Regional Psychoneurological Dispensary, Roshchino, Leningradskaya Oblast'
  - Arkhangelsk Regional Clinical Mental Hospital, Arkhangelsk
  - GUZ Engels Psychiatric Hospital, Engel's
  - Moscow Scientific Research Institute of Psychiatry, Moscow
  - Clinic named after professor Yu. N. Kasatkin FGBOU DPO RMANPO Minzdrava Rossii, Moscow
  - Nizhny Novgorod Region State Institution Of Healthcare Clinical Psychiatric Hospital 1 Of Nizhny ..., Nizhny Novgorod
  - Rostov State Medical University of the Minzdravsotsrazvitiya of Russia, Rostov-on-Don
  - LLC Medical Center Nova Vita, Rostov-on-Don
  - St. Nicolas State Psychiatric Hospital, Saint Petersburg
  - Hospital OrKli , LLC, Saint Petersburg
  - LLC Astarta, Saint Petersburg
  - Saratov State Medical University, Saratov
  - State Budgetery Educational Institution Of Higher Professional Education Smolensk State Medical U..., Smolensk
  - Yaroslavl Regional Clinical Psychiatry Hospital, Yaroslavl
- Slovakia (6):
  - Psychiatricka ambulancia, MENTUM, s.r.o., Bratislava
  - Epamed, S.R.O, Košice
  - Psycholine S.R.O., Rimavská Sobota
  - Crystal Comfort, s.r.o., Vranov Nad Topou
  - BONA MEDIC s.r.o., Zlaté Moravce
  - Psychiatricka Ambulancia, Zlaté Moravce
- Spain (4):
  - Hospital Universitario Fundacion Alcorcon, Alcorcón, Madrid
  - Centro De Salud Mental La Corredoria, Oviedo, Principality of Asturias
  - Hospital De La Santa Creu I Sant Pau, Barcelona
  - Hospital Psiquiatric de Palma de Mallorca, Palma de Mallorca
- Sweden (5):
  - Smaert & Psykiatricentrum Malmoe, Malmo, Skåne County
  - Affecta Psyikiatri AB, Halmstad
  - ProbarE i Lund, Lund
  - ONE LIFETIME Lakarmottagning, Skövde
  - ProbarE, Stockholm
- Ukraine (11):
  - Communal Non-commercial Enterprise Cherkasy regional psychiatric hospital of Cherkasy regional co..., Smila, Cherkasy Oblast
  - Communal Non-Commercial Enterprise of Kharkiv Regional Council Regional clinical psychiatric hosp..., Kharkiv, Kharkivska
  - Municipal Non-profit Enterprise Odesa Regional Psychiatric Hospital No.2 of Odesa Regional Council, Kominternivskyy, Odesa Oblast
  - CI of KRC Regional psychiatric and narcological medical association, Hlevakha
  - Ivano-Frankivsk Oblast neuropsychiatric hospital No. 3, Ivano-Frankivsk
  - Academy of Medical Sciences of Ukraine - Institute of Neurology, Psychiatry and Narcology, Kharkiv
  - SI INPN Namsu, Kharkiv
  - Lviv Regional State Clinical Psychiatric Hospital, Lviv Danylo Galytsky National Medical University, Lviv
  - Odessa Regional Medical Centre of Mental Health, Odesa
  - Ukrainian Medical Stomatological Academy, Chair Of Psychiatry, Narcology And Medical Psychology B..., Poltava
  - Vinnitsa National Medical University, Vinnitsa

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Gill H, McIntyre RS, Christensen MC. Analysis of reward behavior in patients with MDD and partial response to SSRI therapy treated with vortioxetine versus desvenlafaxine: Experience with the Effort-Expenditure for Rewards Task (EEfRT) in the VIVRE study. J Affect Disord. 2025 Nov 1;388:119563. doi: 10.1016/j.jad.2025.119563. Epub 2025 May 31. PMID 40456468
- [Derived] McIntyre RS, Florea I, Pedersen MM, Christensen MC. Head-To-Head Comparison of Vortioxetine Versus Desvenlafaxine in Patients With Major Depressive Disorder With Partial Response to SSRI Therapy: Results of the VIVRE Study. J Clin Psychiatry. 2023 May 22;84(4):23m14780. doi: 10.4088/JCP.23m14780. PMID 37227402